CLINICAL TRIAL: NCT07207005
Title: Comparison of Wear Between Two Dual-mobility Acetabular Cups in Patients Undergoing Total Hip Arthroplasty
Acronym: CUPUSURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A02615-42
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hip Arthroplasty Replacement
Keywords: Hip Arthroplasty Insert

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Highly cross-linked PE (Experimental): The hip prosthesis will be a MOBILIT acetabular cup (Corin), MEIJE femoral stem (Corin), 28 mm diameter metal ball (Corin), and mobile cup (Corin) made of highly cross-linked PE doped with vitamin E (ECIMA, Corin).
  Interventions: Device: ECIMA CORIN
- Conventional PE (Active Comparator): The hip prosthesis will be a MOBILIT (Corin) acetabular prosthesis, MEIJE (Corin) femoral stem, 28 mm diameter metal ball (Corin), and mobile cup (Corin) in conventional PE.
  Interventions: Device: CORIN

INTERVENTIONS:
Device: ECIMA CORIN — Mobile cup (Corin) made of highly cross-linked PE doped with vitamin E (ECIMA, Corin).
  Arms: Highly cross-linked PE
Device: CORIN — Mobile cupule (Corin) is made of conventional PE
  Arms: Conventional PE

SUMMARY:
In 2022, data from the UK's National Joint Registry (NJR) and the American Joint Replacement Registry (AJRR) indicated that Total Hip Replacement (THR) is the most commonly performed orthopaedic joint surgery.

The NJR has observed that between 10 and 20% of hip implants require revision within the first 10 years. The main reasons for these revisions include implant fractures, joint incompatibility, aseptic loosening, dislocation and wear of the polyethylene (PE) insert.

To address this problem, highly cross-linked polyethylene (HXLPE) inserts have been developed. Cross-linking helps to limit wear on polyethylene prostheses in total hip arthroplasty. However, there are concerns about the loss of elasticity of HXLPE and oxidation after implantation.

A new generation of inserts based on highly cross-linked polyethylene (irradiation dose ≥100 Kgy), enriched with vitamin E, has been developed. This PE, called ECIMA, was developed to maintain mechanical properties, minimise PE wear and improve long-term oxidation resistance.

In the HAS evaluation report on highly cross-linked polyethylene inserts dated 24 January 2023, data from the literature show less wear of highly cross-linked polyethylene compared to conventional polyethylene.

Nevertheless, the use of highly cross-linked polyethylene is not yet the gold standard. Furthermore, the data in the literature mainly concern single-mobility cups but not double-mobility cups. Finally, new imaging protocols now make it possible to assess the wear of prosthesis materials more accurately.

In this context, it seems appropriate to conduct a French study comparing double-mobility cups containing highly cross-linked polyethylene or conventional polyethylene inserts.

DETAILED DESCRIPTION:
In 2022, data from the UK's National Joint Registry (NJR) and the American Joint Replacement Registry (AJRR) indicated that total hip arthroplasty or Total Hip Replacement (THR) is the most commonly performed orthopaedic joint surgery.

THR involves replacing worn and damaged areas of cartilage in the hip with artificial parts of similar shape and size. A total hip replacement consists of two parts:

* A part designed to replace the head of the femur: a spherical prosthesis mounted on a stem that is inserted into the femur;
* A part designed to replace the acetabulum: the acetabular cup. There are single-mobility cups and double-mobility cups, where an insert is positioned on the metal head inside a single-mobility cup. Introduced in the 1960s by Sir John Charnley, UHMWPE (Ultra High Molecular Weight Polyethylene) remains the most widely used material for inserts in 2024.

The NJR has observed that between 10 and 20% of hip implants require revision within the first 10 years. The main reasons for these revisions include implant fractures, joint incompatibility, aseptic loosening, dislocation and wear of the polyethylene (PE) insert.

To address this problem, highly cross-linked polyethylene (HXLPE) inserts have been developed. Cross-linking helps to limit wear on polyethylene prostheses in total hip arthroplasty. However, there are concerns about the loss of elasticity of HXLPE and oxidation after implantation.

A new generation of inserts based on highly cross-linked polyethylene (irradiation dose ≥100 Kgy), enriched with vitamin E, has been developed. This PE, called ECIMA, was developed to maintain mechanical properties, minimise PE wear and improve long-term oxidation resistance.

In the HAS evaluation report on highly cross-linked polyethylene inserts dated 24 January 2023, data from the literature show less wear of highly cross-linked polyethylene compared to conventional polyethylene.

Nevertheless, the use of highly cross-linked polyethylene is not yet the gold standard. Furthermore, the data in the literature mainly concern single-mobility cups but not double-mobility cups. Finally, new imaging protocols now make it possible to assess the wear of prosthesis materials more accurately.

In this context, it seems appropriate to conduct a French study comparing double-mobility cups containing highly cross-linked polyethylene or conventional polyethylene inserts.

In the principal investigator's current practice, prostheses with conventional PE inserts are used for patients aged 70 or over, while prostheses with highly cross-linked PE inserts are used for patients under 70. However, this age-based choice is modulated favourably or unfavourably by two other parameters: the patient's medical history and general condition.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged between 55 and 80.
* Patient with a life expectancy > 5 years at the time of inclusion.
* Patient scheduled to undergo primary total hip arthroplasty with a dual-mobility cup prosthesis.
* Patient affiliated with or beneficiary of a social security scheme.
* Patient who speaks French and has signed an informed consent form.

Exclusion Criteria:

* Patients with a contraindication mentioned in the instructions for use of the medical device under investigation
* Patients with an ASA score of 4
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision
* Patients participating in another clinical study whose objectives could interfere with this study

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2036-08-31 (Estimated); Study Completion 2036-08-31 (Estimated)

PRIMARY OUTCOMES:
Femoral head penetration into the acetabulum | Year 5
  Femoral head penetration into the acetabulum will be mesaured in mm/year, based on a hip X-ray and PolyWare® software, Rev 8, Draftware Inc, North Webster, IN, USA

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France, France

IPD SHARING:
Plan to Share IPD: No